CLINICAL TRIAL: NCT01170546
Title: Effects of Hamstring Training in Different Modes on Stabilizing Knee Joints With Anterior Drawer Laxity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Physical Education College (Other)
Responsible Party: Human Subject Committee, Taipei Physical Education College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 950101002
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Results first posted 2010-09-06 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-09

CONDITIONS: Knee Instability
Keywords: anterior cruciate ligament; agility; knee stability; hamstring; knee internal rotator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- KLCIR (Experimental): plate-loaded kneeling leg curl with internal rotation
  Interventions: Other: plate-loaded kneeling leg curl with internal rotation
- SP (Squat Press) (Experimental): plate-loaded squat press
  Interventions: Other: plate-loaded squat press
- KLC (Kneeling Leg Curl) (Experimental): plate-loaded kneeling leg curl
  Interventions: Other: plate-loaded kneeling leg curl

INTERVENTIONS:
Other: plate-loaded kneeling leg curl with internal rotation — The participant was instructed to point toes toward medial side as knee flexing. This is an open-kinetic chain (OKC) exercise and medial hamstring was emphasized.
  Arms: KLCIR
Other: plate-loaded squat press — The subject was instructed to position his back properly against the backrest on a machine, with the feet slightly apart. He was instructed to place his feet higher on the foot plate and draw his two knees as close as possible while the knees flexed so that medial hamstring would supposedly bear more tension in the course of knee flexion. This is a closed-kinetic chain (CKC) exercise and was expected to strengthen the quadriceps and hamstring with medial hamstring emphasized.
  Other Names: angled leg presses
  Arms: SP (Squat Press)
Other: plate-loaded kneeling leg curl — An open-kinetic chain (OKC) exercise was intended to strengthen the hamstring muscle without lateralization emphasized.
  Arms: KLC (Kneeling Leg Curl)

SUMMARY:
Question: To investigate how different modes of thigh muscles strengthening exercises emphasizing the knee internal rotators can be as effective as possible in improving the static stability and agility of the knees with anterior drawer laxity.

Design: Randomized controlled clinical trial.

Participants and Interventions:

Young men with anterior drawer laxity of the knee were randomly assigned to three experimental groups in different strengthening modes: plate-loaded squat press (SP), plate-loaded kneeling leg curl with internal rotation (KLCIR), and kneeling leg curl (KLC). The control group with stable knees received no training.

Outcome measures: static and dynamic knee stability, isokinetic strength. The purpose of this paper was to find out an optimal solution to the enhancement of the static and dynamic knee stability to a great extent.

Key words: anterior cruciate ligament; agility; knee stability; hamstring; knee internal rotator

DETAILED DESCRIPTION:
INTRODUCTION Anterior cruciate ligament (ACL) injuries are commonly seen among athletes, which eventually makes more or less devastating impacts on their performances. Although ACL injuries may result from the knee collision, 70% of them are due to noncontact movements, including abrupt brakes, changing directions at high speed (i.e. sidestep cuttings and crossover cuttings). In doing so, one must at first have his or her axial foot fixed on the ground to absorb the momentum oriented from the original direction. Insufficient eccentric muscles or ligament strength are likely to trigger muscle and ligament injuries.

It is generally agreed that the risk of ligament injuries can be reduced by strengthening a specific muscle group by which the dynamic stability of the joint is able to be enhanced and the static stability provided by the ligament can also be compensated. Traditionally, the strengthening exercise of ACL rehabilitation has been putting an emphasis on the hamstring and quadriceps with an attempt to decrease the anterior drawer instability as well as the shearing force of ACL. Nonetheless, from the aforementioned pathomechanism of ACL injuries, the knee rotators should be valued as they are supposed to . The internal rotators of the knee joint (semitendinosus, semimembranosus and gracilis) are highly related to ACL injuries5. However, the knee rotator strength is often neglected and even sacrificed as an autograft for the ACL reconstruction .

Modifications can be made in progressive resistance exercise for strengthening knee internal rotators. In this current study, 20 subjects with anterior drawer laxity were randomly assigned to three groups adopting different training modes: plate-loaded squat press (SP), plate-loaded kneeling leg curl with internal rotation (KLCIR), and plate-loaded kneeling leg curl (KLC). Static stability, dynamic stability, and isokinetic strength were measured. The purpose of this paper was to find out an optimal solution to the enhancement of the static and dynamic knee stability to a great extent.

MATERIALS AND METHODS Subjects The research program was approved by the Human Subject Committee in Taipei Physical Education College. Knee joint laxity was surveyed by a KT-2000 test (MED Metric Co., San Diego, USA) in the Department of Physical Education and Health at Taipei Physical Education College. The anterior drawer laxity of the knee joint in this study was defined as anterior displacement over 3 mm discrepancy between bilateral knee joints by a KT-2000 test under 20-pound force. According to this criterion, Dale M. et al. demonstrated that 85% (33/39) of this population have complete ACL tears and 15% (6/39) have partial tear. One hundred and seventy-three students were tested and 30 met the criterion, including 22 males and 8 females, although no obvious trauma history was available in some of them. Two males were excluded due to other causes that might affect muscle strength or knee stability such as lower limbs fracture and arthritis. Besides, eight female students were eliminated to avoid possible gender difference. Twenty male students were included in the experimental group. Another 8 male students with stable knees without any medical history of knee injuries were included in the control group. The participants in both experimental and control groups lived a sedentary lifestyle. Stable knees were defined as a discrepancy less than 1.5mm between bilateral knees by a KT-2000 test under 20-pound force.

Flow Path Twenty subjects in the experimental group were randomly assigned into three groups: SP (n=7), KLCIR (n=7) and KLC (n=6). Eight control subjects neither received any training nor was engaged in body-building on their own during the training period. Every subject was asked to fill in basic information, including age, body height, and body weight. Before the experiments, the flow path was explained to each subject who had already signed an informed-consent form.

The experimental procedure was divided into three phases. The first and the third phases were the tests before and after training respectively, including KT-2000, agility, and isokinetic strength assessment. The second phase was the training phase.

Static Stability (Laxity) The KT-2000 knee ligament arthrometer (MED Metric Co., San Diego, USA) is designed to assess the anterior drawer laxity of the knee joint. The discrepancy of anterior displacement between the sound side and the lesion side had been reported and applied in evaluating the static stability of the knee, and it was also used as one of the references for the ACL reconstruction surgery. In this current study, a discrepancy less than 1.5mm was normally accepted when 20-pound anterior traction force was exerted on the tibia with the knee joint in 20° flexion. In contrast, ACL laxity was defined as a discrepancy over 3mm, which was highly related to ACL injury.

Dynamic Stability (Agility) Dynamic knee stability was assessed by agility, which was measured by a 6-meter left-and-right shuttle run. A good dynamic knee stability is necessary for changing the movement direction. Each subject started running from the midline to the left terminal and then stepped on the square with his left foot. Then, the subject used the left leg as the axis and turned around to the right side. The subject then ran to the right terminal. Once the front foot was crossing the midline, this was the first round for testing the agility of left knee. The subject kept running to the right terminal without stopping on the midline, stepping on the square with his right foot, turning around to the left side, and running toward the left terminal. This was the first round of right knee test as the subject's front foot crossed the midline. Whenever the front foot crossed the midline, a timer was clocked. The time interval in seconds between the 1st and the 2nd time clocked was the 1st measure of the left knee agility, and the time interval between the 2nd and the 3rd was the 1st measure of the right knee agility, and so forth. There were five-round tests for the agility of right and left knees respectively. Three raters were assigned respectively at the midline, right and left terminals. Single-blind method was adopted. That is, all the three raters did not know which group the subject was assigned to. The square at the right or left terminal ends was 10 inches wide and 3 meters away from the midline. It would be recognized as a qualified round if the plantar surface of the foot ever contacted any part of the square; otherwise, the subject would be asked to repeat the whole set consisting of five rounds. Three sets were collected and averaged. The rest interval between each set should be long enough for the examinee to feel relaxed before the next set. The subject was asked to run as fast as possible. The average time difference of 3 sets between the affected and the sound side was regarded as the dynamic stability of the affected side. The greater the difference was, the poorer the dynamic stability or the agility would be. A practice session was given prior to the actual beginning of the study to avoid learning effect.

Prior to the study, intrarater test-retest reliability was established. Nine subjects, including four in the experimental groups and five in the control group, took the agility exam twice in separated days. The intraclass correlation coefficient was 0.78.

Isokinetic Strength Cybex NORM (Cybex International, Inc, Ronkonkoma, New York, U.S.A.) was employed to evaluate isokinetic muscle strength before and after training. Tests were conducted in two different motion modes which included the flexor/extensor and the internal /external rotator. In the former, the range of motion was set in the range of 0-90°. Maximal concentric force had been performed for five times at the angular velocity of 60°, 120° and 180° per second, respectively. Peak torque was taken to represent muscle strength. Only smooth and similar curves with a peak torque which was no less than 90% of the maximum would be taken. The assessment of isokinetic strength of internal/external rotator was generally similar to flexor/extensor. The ankle joint was fixed into 30° dorsiflexion with an air-stirrup ankle brace (Aircast, Summit, NJ) to limit unnecessary inversion/eversion movement, which might affect measurement of knee joint rotation. In addition, the knee and hip joints were kept in 90°, and the range of motion of knee rotation was set in the range between 25° internally and 35° externally.

Training Modes Three training modes were chosen. (Ⅰ) SP (or called angled leg presses); (Ⅱ) KLCIR; (Ⅲ) KLC. The training phase had been lasting for 6 weeks in which none dropped out. Each subject had to accomplish three training workouts weekly under supervision by licensed athletic trainers. A workout contained five sets for each lower limb, which were composed of 20 (repetitions)×60% (1RM), 15×65% , 12×70% , 8×75% and 20×60% with a two-minute resting interval between each set. During the six-week rehabilitation course, they were not allowed to involve in any other regular fitness activities or sports.

Data Analysis Data are expressed as mean±SEM. SPSS version 12.0 Windows was used for statistic analysis. Nonparametric analysis, including Kruskal-Wallis Test, Wilcoxon Test and Mann-Whitney test, was applied. Significance was defined as P<0.05. Intrarater reliability was assessed with intraclass correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* The anterior drawer laxity of the knee joint in this study was defined as anterior displacement over 3 mm discrepancy between bilateral knee joints by a KT-2000 test under 20-pound force.

Exclusion Criteria:

* anterior displacement less than 3 mm discrepancy between bilateral knee joints by a KT-2000 test under 20-pound force.

Ages: 15 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2006-01; Primary Completion 2007-01 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Wei Chou, Principal Investigator — Department of Physical Medicine and Rehabilitation, Chang Gung Memorial Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Chang Gung Memorial Hospital, Taipei, Taiwan, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Knee joint laxity was surveyed by a KT-2000 test during 2006, Feb and 2006, March. The anterior drawer laxity of the knee joint was defined as anterior displacement over 3 mm discrepancy between bilateral knee joints by a KT-2000 test under 20-pound force.
Pre-assignment Details: One hundred and seventy-three students were tested and 30 met the criterion, including 22 males and 8 females. Two males were excluded due to other causes that might affect muscle strength or knee stability such as lower limbs fracture and arthritis. Besides, eight female students were eliminated to avoid possible gender difference.
Groups:
- KLC ( Kneeling Leg Curl): plate-loaded kneeling leg curl
- Control: Control group
Period: Overall Study
Arm/Group | KLCIR | SP (Squat Press) | KLC ( Kneeling Leg Curl) | Control
Started | 7 | 7 | 6 | 8
Completed | 7 | 7 | 6 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KLCIR | SP (Squat Press) | KLC ( Kneeling Leg Curl) | Control | Total
Number analyzed (Participants) | 7 | 7 | 6 | 8 | 28
Age Categorical [Number; unit: participants]
  Between 18 and 25 years | 7 | 7 | 6 | 8 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 20.6 (0.42) | 20.3 (0.49) | 20.3 (0.8) | 21.5 (0.78) | 20.7 (0.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 7 | 7 | 6 | 8 | 28
Region of Enrollment [Number; unit: participants]
  Taiwan | 7 | 7 | 6 | 8 | 28

OUTCOME MEASURES:

1. Primary Outcome: Static Knee Stability
Description: The KT-2000 knee ligament arthrometer (MED Metric Co., San Diego, USA) is designed to assess the anterior drawer laxity of the knee joint. The discrepancy of anterior displacement between the sound side and the lesion side is applied in evaluating the static stability of the knee.
Time Frame: one year
Reporting Status: Not Posted, anticipated posting 2010-12
Measure: Mean (Standard Error); unit: mm

2. Primary Outcome: Agility
Description: shuttle run agility test
Time Frame: one year
Reporting Status: Not Posted, anticipated posting 2010-12
Measure: Mean (Standard Deviation); unit: sec.

3. Primary Outcome: Isokinetic Strength
Description: Cybex NORM (Cybex International, Inc, Ronkonkoma, New York, U.S.A.) was employed to evaluate isokinetic muscle strength before and after training.
Time Frame: one year
Reporting Status: Not Posted, anticipated posting 2010-12
Measure: Mean (Standard Error); unit: ° / sec

4. Primary Outcome: Age
Time Frame: before training
Measure: Mean (Standard Deviation); unit: year
Arm/Group | KLCIR | SP (Squat Press) | KLC ( Kneeling Leg Curl) | Control
Number analyzed (Participants) | 7 | 7 | 6 | 8
year | 20.6 (0.42) | 20.3 (0.49) | 20.3 (0.8) | 21.5 (0.78)

ADVERSE EVENTS:
Arm/Group | KLCIR | SP (Squat Press) | KLC ( Kneeling Leg Curl) | Control
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/8

LIMITATIONS AND CAVEATS:
small size, participant: not real ACL-injured patient but knee with anterior laxity instead

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No